CLINICAL TRIAL: NCT05847660
Title: A Randomized Controlled Study of Progesterone Primed Ovarian Stimulation Protocol Versus Antagonist Protocol for PCO Patients in Intracytoplasmic Sperm Injection Cycles
Brief Title: Progesterone Primed Ovarian Stimulation Protocol Versus Antagonist Protocol for PCO Patient
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, rehab abdelhamid aboshama, associate professor of obstetrics and gynecology, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: D 319
Record Dates: First submitted 2023-04-27; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Ovary Syndrome; Infertility; IVF
Keywords: Polycystic ovary disease; ICSI; progesterone; antagonist protocol
MeSH Terms: conditions — Polycystic Ovary Syndrome; Infertility | interventions — Dydrogesterone; cetrorelix

STUDY DESIGN:
Intervention Model Description: this is a randomized controlled non-blinded study. it will include 210 pt all of them PCO pt with infertility
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Progesterone primed ovarian stimulation protocol. (Active Comparator): Group (A): Women in progesterone primed (PPOS) will be prescribed a 30 mg oral dose of dydrogesterone (Duphaston, Abbott, Egypt) from the 2nd day of the cycle and continued until the triggering day. Vaginal sonography will be done for all patients since 6th day of the cycle.
  Interventions: Drug: Progesterone antagonist
- conventional antagonist protocol. (Active Comparator): Group (B): Women in the antagonist group will be monitored by transvaginal ultrasonography till the size of dominant follicles reached to 12-13 mm, 0.25 mg of Cetrotide (Merck-Serono, Germany) will be injected subcutaneously daily and continued until triggering day, follow up for all patients in both groups by transvaginal ultrasound every other day.
  Interventions: Drug: conventional antagonist protocol

INTERVENTIONS:
Drug: Progesterone antagonist — Group (A): Women in progesterone primed (PPOS) will prescribed 30 mg oral dose of dydrogesterone (duphaston, Abbott, Egypt) from the 2nd day of the cycle and continued until triggering day. Vaginal sonography will be done for all patients since the 6th day of the cycle.
  Other Names: duphaston
  Arms: Progesterone primed ovarian stimulation protocol.
Drug: conventional antagonist protocol — Group (B): Women in the antagonist group will be monitored by transvaginal ultrasonography till the size of dominant follicles reached to 12-13 mm, 0.25 mg of cetrotide (Merck-Serono ,Germany) will be injected subcutaneously daily and continued until triggering day, follow up for all patients in both groups by transvaginal ultrasound every other day.
  Other Names: 0.25 mg of cetrotide
  Arms: conventional antagonist protocol.

SUMMARY:
this study is designed to compare the Progesterone primed ovarian stimulation protocol versus the antagonist protocol as a method to stimulate PCO patients in ICSI cycles to decrease cost and decrease OHSS.

DETAILED DESCRIPTION:
A Randomized controlled, non-blinded study (parallel-group study with 1:1 randomization) will be conducted at a Specialized Authorized IVF unit starting from January 2023 till completing the sample size. Randomization will be generated by a computer and held with one of the experimenters, and (n) of the black and red cards will be used for allocation concealment.

Participants: All PCO patients will be given informed consent about the study aims and written consent will be taken at the first visit to the infertility clinic of the Specialized Authorized IVF unit.

Patients will be categorized as (Group A) Progesterone primed ovarian stimulation protocol. (Group B) conventional antagonist protocol.

ELIGIBILITY:
Inclusion Criteria:

- 1. PCO patients based on Rotterdam criteria (2003), including polycystic ovaries, oligo-anovulation, as well as the biochemical or clinical signs of hyperandrogenism (Rotterdam et al, 2003).

2. Age less than 40 years old. 3. Primary infertility for 2 years and secondary infertility for 1 year.

Exclusion Criteria:

- Non-PCO patients as:

* Congenital adrenal hyperplasia
* Hyperprolactinemia.
* Recurrent implantation failure.
* Hydrosalpinx.
* Uterine pathology.
* Uncontrolled medical disorder eg DM, HTN
* Male factor infertility.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 210 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-07-01 (Estimated)

PRIMARY OUTCOMES:
The number of oocytes retrieved per patient | 12 months
  The number of oocyte retieved by ovum pick up after controlled ovarien stimulation
The number of MII oocytes/per patient | 12 months
  the grade of maturity of oocyte under microscope
The fertilization rate/per patient. | 12 months
  The number of fertilized oocyte by sperm
Number of frozen embryos/per patient | 12 month
  the number of embryo frozen

SECONDARY OUTCOMES:
Incidence of early OHSS yes /no | 12 months
  size of th overies , presence of ascitis , pain and
Pregnancy outcomes | 12 months
  1. Chemical pregnancy will be determined by serum β hCG > 50 IU/L two weeks after ET.
  2. In addition, clinical pregnancy will be confirmed by detecting fetal heartbeats 2 weeks following the positive β hCG.